CLINICAL TRIAL: NCT04243382
Title: Treatment of Children With Autistic Spectrum Disorder With Autologous Umbilical Cord Blood, a Pilot Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Omer Bar-Yosef, M.D.-Ph.D. Peadiatric Neurology and Child Development. The Edmond and Lily Safra Children's Hospital, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHEBA-18-5105-OBY-CTIL
Record Dates: First submitted 2020-01-15; First posted 2020-01-28 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Autistic Spectrum Disorder
Keywords: Autistic Spectrum Disorder, autologous umblical cord blood
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomization will be done by external source and the assignment will disclosed to cord bank bank only. They will produce either a cord blood or placebo unit which will be completely covered. Each unit will have its own index number that will be documented by the research coordinator. Neither the researcher or the family will know the nature of the unit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Experimental): Autologous umbilical cord blood transfusion Single dose of an Autologous umbilical cord blood transfusion
  Interventions: Biological: Autologous umbilical cord blood
- group 2 (Experimental): The placebo product will consist of the standard ingredients of the acellular content of the UCB unit. It will consist of 20 ml Dextran (Plander 40.000 - 50g/500ml, solution for infusion) and 20 ml of human Albumin 5% (solution for infusion). The volume of placebo product will be 40 ml,
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Autologous umbilical cord blood — Single infusion of autologous umbilical cord blood cells
  Arms: group 1
Biological: Placebo — Placebo
  Arms: group 2

SUMMARY:
This study is a phase II, prospective, double blind, placebo-controlled study of the efficacy of autologous umbilical cord blood infusion.

The study population will consist of 60 children ages 18 months to 12 years with ASD. The population will be randomly assigned to 2 groups, the study group be treated by cord blood in the beginning of the study and the control group by placebo product.

The study will consist of 4 stages Stage 1: initial assessment by physiotherapist and occupational therapist / treatment by cord blood or placebo / blood work before and after treatment Stage 2: at stage 1 + 6 months assessment by physiotherapist and occupational therapist / cross-over treatment by cord blood or placebo / blood work before and after treatment Stage 4: at stage 1 + 12 months assessment by physiotherapist and occupational therapist The primary outcome is improvement of social communication skills six months after treatment at stage 1

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 1.5 years to ≤ 12 years (11 years, 364 days) at the time of visit 1
* Confirmed clinical DSM-5 diagnosis of Autism Spectrum Disorder using the DSM-5 criteria
* Fragile X testing performed and negative
* Available and qualified umbilical cord blood unit with a minimum banked total nucleated cell dose of ≥ 2 x 10e7 cells/kg
* Stable on current psychiatric medication regimen (dose and dosing schedule) for at least 2 months prior to infusion of study product
* Normal absolute lymphocyte count (≥1500/uL)
* Able to travel to Sheba Medical Center University three times (baseline, 6 and 12 months post-baseline), and parent/guardian is able to participate in interim surveys and interviews monthly
* Parental consent

Exclusion Criteria

* General:

  * Review of medical records indicates ASD diagnosis not likely
  * Known diagnosis of any of the following coexisting psychiatric conditions: depression, bipolar disorder, schizophrenia, obsessive compulsive disorder
  * Screening data suggests that participant would not be able to comply with the requirements of the study procedures, including study outcome measures, as assessed by the study team
  * Family is unwilling or unable to commit to participation in all study-related assessments, including follow up for approximately 12 months
* Genetic:

  * Records indicate that child has a known genetic syndrome such as (but not limited to) Fragile X syndrome, neurofibromatosis, Rett syndrome, tuberous sclerosis, PTEN mutation, cystic fibrosis, muscular dystrophy
  * Known pathogenic copy number variation (CNV) associated with ASD (e.g., 16p11.2, 15q13.2, 2q13.3)
* Infectious:

  * Known active CNS infection
  * Evidence of uncontrolled infection based on records or clinical assessment
  * HIV positivity
* 4 Medical:

  * Known metabolic disorder
  * Known mitochondrial dysfunction
  * History of unstable epilepsy or uncontrolled seizure disorder, Lennox Gastaut syndrome, Dravet syndrome, or other similar epileptic encephalopathy
  * Concurrent genetic or acquired disease or comorbidity(ies) that could require a future stem cell transplant
  * Significant sensory (e.g., blindness, deafness, uncorrected hearing impairment) or motor (e.g., cerebral palsy) impairment
  * Evidence of clinically relevant physical dysmorphology indicative of a genetic syndrome as assessed by the PIs or other investigators, including a medical geneticist and psychiatrists trained in identifying dysmporphic features associated with neurodevelopmental conditions.
* Current/Prior Therapy:

  * History of prior cell therapy
  * Current or prior use of IVIG or other anti-inflammatory medications with the exception of NSAIDs
  * No systemic steroid therapy that has lasted >2 weeks, and no systemic steroids within 3 months prior to enrollment. Topical and inhaled steroids are permitted.

Ages: 18 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2020-02-27 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Improvement of social communication skills | 6 months
  Vineland Adaptive Behavior Scales-Second Edition (VINELAND-II)
Improvement of social communication skills | 6 months
  Pediatric Evaluation of Disability Inventory-Computer Adaptive Test-ASD

SECONDARY OUTCOMES:
Improvement of social communication skills | 6 months
  Theory of Mind Inventory - 2
Functional assessment | 6 months
  Adaptive Behavior Assessment System - Second edition (ABAS-2)

CONTACTS AND LOCATIONS:
Overall Officials: Omer Bar-Yosef, MD.PHD, Principal Investigator — Sheba Medical Center
Locations (1):
- Chaim Seba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Yes
Yes data set of the baseline of the children, the quantity of cord blood transfusion they received and the clinical followup information.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: within 2 years from the end of data collection

REFERENCES:
- [Background] Lai MC, Lombardo MV, Baron-Cohen S. Autism. Lancet. 2014 Mar 8;383(9920):896-910. doi: 10.1016/S0140-6736(13)61539-1. Epub 2013 Sep 26. PMID 24074734
- [Background] Christensen DL, Baio J, Van Naarden Braun K, Bilder D, Charles J, Constantino JN, Daniels J, Durkin MS, Fitzgerald RT, Kurzius-Spencer M, Lee LC, Pettygrove S, Robinson C, Schulz E, Wells C, Wingate MS, Zahorodny W, Yeargin-Allsopp M; Centers for Disease Control and Prevention (CDC). Prevalence and Characteristics of Autism Spectrum Disorder Among Children Aged 8 Years--Autism and Developmental Disabilities Monitoring Network, 11 Sites, United States, 2012. MMWR Surveill Summ. 2016 Apr 1;65(3):1-23. doi: 10.15585/mmwr.ss6503a1. PMID 27031587
- [Background] Prata J, Santos SG, Almeida MI, Coelho R, Barbosa MA. Bridging Autism Spectrum Disorders and Schizophrenia through inflammation and biomarkers - pre-clinical and clinical investigations. J Neuroinflammation. 2017 Sep 4;14(1):179. doi: 10.1186/s12974-017-0938-y. PMID 28870209